CLINICAL TRIAL: NCT06598215
Title: Hybrid Duckett Urethroplasty Versus Modified Single Stage Duckett Uteothroplasty for Management of Proximal Hypospadias: a Randomized Clinical Trial
Brief Title: Hybrid Duckett vs Modified Duckett Urethroplasty for Proximal Hypospadias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammad Gharieb Mohammad Khirallah, professor of pediatric surgery, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35171/12/21
Record Dates: First submitted 2024-08-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Proximal Hypospadias; Modified Duckett Urethroplasty
Keywords: proximal hypospadias; staged repair; Duckett urethroplasty; urethrocutaneous fistula; chodree

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A hybrid Duckett urethroplasty (Active Comparator)
  Interventions: Procedure: Duckett urethroplasty
- group B modified Duckett urethroplasty (Active Comparator)
  Interventions: Procedure: Duckett urethroplasty

INTERVENTIONS:
Procedure: Duckett urethroplasty — hybrid duckett urethroplasty vs modified duckett urethroplasty

SUMMARY:
proximal hypospadias presents a serious anomaly for both infants and their care givers. a variety of techniques were described through decades. None of them is completely curable. hundred of modifications were adopted to the original techniques. during the current study, we will do hybrid Duckett urethroplasty which is a staged procedure and compare it to modified Duckett urethroplasty which is a single stage procedure.

DETAILED DESCRIPTION:
two groups of infants diagnosed with proximal hypospadias will be allocated in two groups. group A will include cases of who will be operated upon using hybrid Duckett urethroplasty. group B will include patients who will be operated upon using modified duckett urethroplasty.

recruitment in either group will be done using sealed envelop method. in group A patient will have a double face Duckett tube which will be transferred to the ventral of the penis. the tube will be secured in place however, no proximal anastomosis with the meatus. the anastomosis will be scheduled six months later. In group B patients a double face Duckett tube will be transferred to the ventral aspect of the penis with completion of the anastomosis with the proximal meatus at the same session. the primary out come will be completion of the procedure and restoration of the urethral continuity. secondary out come will the cosmetic appearance

ELIGIBILITY:
Inclusion Criteria:

* all infants and children with proximal hypospadias

Exclusion Criteria:

* disorders of sex developments
* previous penile surgery
* circumcised children
* crippled penis
* refusal of the plan of the management by the care givers

Ages: 6 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
repair of proximal hypospadias without fistula | six months post operative
  strong strait stream of urine, no fistula formation, no urethral stricture

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Elgharbeya, Egypt

IPD SHARING:
Plan to Share IPD: No
the preoperative photos, operative photos and postoperative photos will be sharable with other researchers